CLINICAL TRIAL: NCT04210648
Title: Effectiveness and Security Testing of a Mobile App for Self-Managing Emotion Dysregulation in a Non-Clinical Population With Borderline Traits: A Randomized Controlled Trial
Brief Title: Effectiveness and Security Testing of a Mobile App for Self-Managing Emotion Dysregulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari del Maresme (Other)
Collaborators: University Ramon Llull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 32-16
Record Dates: First submitted 2019-12-19; First posted 2019-12-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Emotional Dysregulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Those who will use the mobile app
  Interventions: Device: Mobile app
- Non-intervention group (No Intervention): Those who will not use the mobile app

INTERVENTIONS:
Device: Mobile app — Mobile app for self-managing emotional dysregulation
  Arms: Intervention group

SUMMARY:
To assess the effectiveness and security of a mobile App (beta version) for people with borderline traits recruited from a non-clinical population of college students in Barcelona (Spain). The main primary outcome will be the severity of the emotional dysregulation. Forty participants will use the mobile app over 6 months. This group while be compared at post-treatment and at 3-month follow-up with other 40 participants (control group) with any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Borderline traits
* Aged between 18 to 65 years
* College students

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Emotion dysregulation severity | 9-month
  Severity of emotional dysregulation as measured by a single score from the The DERS scale (Difficulties in Emotion Regulation scale) (range: 0-88; the higher the score, the more severe the emotion dysregulation severity).
smartphone addiction | 9-month
  Severity of smartphone addiction as measured by the Spanish version of the The Smartphone Addiction Scale (SAS) (range: 10-60; the higher the score, the more severe the smartphone addiction severity).

IPD SHARING:
Plan to Share IPD: No